CLINICAL TRIAL: NCT07044050
Title: A First-in-human, Open-label, Clinical Study to Assess the Safety, Tolerability, and Activity of OT-C001 (Amplified/Activated Allogenic Natural Killer Cells) in Patients With Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: A First-in-human Study to Assess OT-C001 (Amplified/Activated Allogenic Natural Killer Cells) in Patients With Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emercell SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C00101
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-cell Lymphoma With no Other Specification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Dose Level 1) (Experimental): OT-C001 1 vial, weekly dosing
  Interventions: Biological: allogenic natural killer cells
- Cohort 2 (Dose Level 2) (Experimental): OT-C001 3 vials, weekly dosing
  Interventions: Biological: allogenic natural killer cells
- Cohort -1 (Sub Dose Level) (Experimental): OT-C001 1/3 vial (100M)
  Interventions: Biological: allogenic natural killer cells

INTERVENTIONS:
Biological: allogenic natural killer cells — OT-C001 will be administered by IV infusion weekly for at least 3 doses.
  Other Names: OT-C001; NK-001

SUMMARY:
The goal of this clinical trial is to learn the safety of OT-C001 and decide a good dose in treating relapsed or refractory diffuse large B-cell lymphoma patients. It will also learn about the preliminary activity of OT-C001.

Participants will:

Receive a short course of chemotherapy before OT-C001 treatment. During the study treatment, participants will recieve weekly dose of OT-C001 for 3 or 6 weeks. During the study period, participants will also receive another two drugs, rituximab and IL-2, to support OT-C001 treatment.

Participants need to visit the clinic or may be hospitalized according to the study plan.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* histologically confirmed diagnosis of R/R DLBCL-NOS without further standard treatment options including those relapsing after or ineligible for CAR T-cell therapy
* with evaluable disease
* with adequate biological parameters at baseline
* ECOG performance status ≤1
* life expectancy >3 months as assessed by the investigator

Exclusion Criteria:

* Receive concomitantly any antitumor-directed drug therapy
* Any vaccination with live virus vaccines before or during treatment
* With severe atopic predisposition who need a treatment with monoclonal antibodies, allergen immunotherapy, or long-term systemic corticosteroids
* Major surgery within 3 weeks
* With rapidly progressing disease that includes massive uncontrolled pleural, pericardial, or peritoneal effusions, pulmonary lymphangitis, and over 50% liver involvement
* Ongoing immune-related tocivities or adverse events grade >1 not resolved from previous therapies except vitiligo, stable neuropathy up to grade 2, hair loss, and stable endocrinopathies with substitutive hormone therapy
* Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy within the last 12 months
* Primary or secondary immune deficiency
* Active and uncontrolled infections requiring intravenous antibiotic or antiviral treatment
* Seropositive (except after vaccination or confirmed cure for hepatitis) for HIV, HBV, or HCV
* Clinically significant cardiac disease including heart failure, uncontrolled hypertension, pre-existing arrhythmia, uncontrolled angina pectoris, or myocardial infarction within 12 months
* Dementia or altered mental status that would prohibit informed consent
* Other malignancy within the last 3 years except adequately treated nonmelanoma skin cancer, in situ carcinoma of the uterine cervix, or myelodysplastic syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and clinically significant findings on clinical laboratory tests, performance status, vital signs, ECGs, and physical examinations. | All assessments will be conducted from first study treatment administration through the End of Treatment or Early Termination Visit (scheduled within 14 days after the last dose).

SECONDARY OUTCOMES:
Antitumor activity characterized by objective response rate per Lugano criteria. | Tumor will be assessed at the end treatment cycles (3 and 6 weeks after the first dose), and every 12 weeks afterwards for up to of 2 years until progression of disease or starting new anti-cancer treatments.

OTHER OUTCOMES:
Duration of OT-C001 persistence after administering OT-C001. | From baseline (before lymphodepletion) to end of study treatment (within 14 days after the last dose of OT-C001).
Changes in serum cytokine levels | From baseline (before lymphodepletion) to end of study treatment (within 14 days after the last dose of OT-C001)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Herrera, Study Chair — Emercell SAS
Locations (1):
- Saint-Eloi Hospital, Montpellier, France